CLINICAL TRIAL: NCT05068986
Title: Asthma Education and Its Impact on Emergency Department Visits by Asthmatic Children
Brief Title: Asthma Education and Emergency Department Visits by Asthmatic Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AinShamsUISA
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: The Frequency of ER Visits in Asthmatic Children
Keywords: asthma, pediatric, education
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm intervention (Other)
  Interventions: Behavioral: Asthma education

INTERVENTIONS:
Behavioral: Asthma education — All the study participants were subjected to an educational asthma program for 3 months for providing parents and children with information and skills to manage their asthma ,which was presented from the the first session, through providing a written asthma action plan, information about avoiding triggers, training in the correct use of medicines, including inhaler technique, information and support to maximize adherence . All patients were followed up by a phone call every 2 weeks and follow up visit monthly to confirm compliance to the educational program

SUMMARY:
This study will be conducted to evaluate the effects of an educational asthma program on the frequency of emergency department visits and identifying factors associated with frequent emergency department visits by asthmatic children and determine its effect on asthma severity and quality of life among asthmatic children and their caregivers.

DETAILED DESCRIPTION:
This one-arm interventional clinical trial study will be conducted at pediatric chest clinics and the emergency department of the children's hospital of Ain Shams University located in Cairo during the period from September 2021 to the end of December 2021.

The study will be conducted on 30 asthmatic pediatric patients aged from 1-15 years old with documented asthma diagnoses (intermittent wheezes, breathlessness, dry cough, etc)

Inclusion criteria:

: Objective asthma diagnostic testing consists of 2 components: (1) demonstration of airway obstruction and (2) documentation of variability in the degree of obstruction.

Exclusion criteria:

1. Underlying chronic lung diseases like: (Cystic fibrosis, tuberculosis, childhood interstitial lung diseases).
2. Asthmatic patients with major systemic illness (diabetes, chronic renal failure, chronic liver disease).

All the study participants will be subjected to an educational asthma program for 3 months to provide parents and children with information and skills to manage their asthma, through avoiding triggers, training in the correct use of medicines, including inhaler technique, information, and support to maximize adherence. All patients will be followed up by a phone call every 2 weeks and a follow-up visit monthly to confirm compliance with the educational program.

ELIGIBILITY:
Inclusion Criteria:

* Children with a documented asthma diagnosis Children aged from 1 to 15 years

Exclusion Criteria:

* Children with underlying chronic lung diseases

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2021-09-26 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
The emergency room visits frequency | 2 months
  to reduce the number of ER visits

CONTACTS AND LOCATIONS:
Locations (1):
- Children hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No